CLINICAL TRIAL: NCT05361356
Title: Spectral CT Clinical Trial
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Investigational product had been released in NMPA, Sponsor decided to terminate the study aligned with investigator.
Sponsor: Philips (China) Investment CO., LTD (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PD_CT_Hawk_2021_11257
Record Dates: First submitted 2022-03-16; First posted 2022-05-04 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2023-04

CONDITIONS: Adult ALL
Keywords: CT scanning, image assessment
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental group, all volunteer will be scanned. (Experimental): All participation accept Spectral CT scanning; No group;
  Interventions: Radiation: Spectral CT scanning

INTERVENTIONS:
Radiation: Spectral CT scanning — Volunteer accept spectral CT scanning

SUMMARY:
The objective of this clinical trial was to evaluate the efficacy, ease of operation, stability, and safety of Spectral CT as expected.

DETAILED DESCRIPTION:
Under the premise of protecting subjects and ensuring the scientific nature of this clinical trial, Spectral CT was evaluated for its effectiveness, convenience, stability and safety under normal conditions by collecting clinical cases.

ELIGIBILITY:
Inclusion Criteria:

* Volunteers (ages 18 to 75);
* Negative pregnancy tests for women of childbearing age;
* Agree to participate in the clinical trial and sign the subject informed consent form;
* Enhanced scan requires laboratory evidence of normal renal function.

Exclusion Criteria:

* The body cannot comply with CT examination;
* Pregnant and lactating women;
* Claustrophobia;
* People who are not suitable for enhanced scanning with iodine contrast agent (previous severe heart failure and hyperthyroidism, iodine contrast agent allergy and susceptibility);
* Patients deemed unsuitable for participation in this clinical trial by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2022-03-10 (Actual); Primary Completion 2022-10-19 (Actual); Study Completion 2023-02-27 (Actual)

PRIMARY OUTCOMES:
Excellent and good rate of clinical imaging (score≥3） | through study completion, an average of 1 year
  Rated items 5 points Excellent image quality for diagnostic purposes, very satisfactory 4 points good image quality, can be used for diagnosis, satisfactory 3 points Image quality defects, do not affect the diagnosis, general 2. Unsatisfactory image quality, affecting diagnosis Poor image quality, undiagnosable, unsatisfactory

SECONDARY OUTCOMES:
Common functions assessment | through study completion, an average of 1 year
  Common function evaluation items inclduing:The exposure function; Bed body moving; Microphone intercom function; Image post-processing function; Data storage management. With Satisfied, normal, Not Satisfied
Convenience evaluation assessment | through study completion, an average of 1 year
  Convenience function evaluation items inclduing:Laser positioning lamp Breathing navigation Control buttons The clinical interface friendliness of postprocessing software The post-processing software is convenient for clinical use and operation. With Satisfied, normal, Not Satisfied
Machine function and stability assessment | through study completion, an average of 1 year
  Machine function and stability evaluation items inclduing:workflow Image display and transmission Failed to start system Unexpected system shutdown Abnormal termination during the scan Unable to expose during scan. With Satisfied, normal, Not Satisfied
Adverse events and serious adverse events | through study completion, an average of 1 year
  Adverse events and serious adverse events during the test were collected to evaluate the safety of the product.

CONTACTS AND LOCATIONS:
Overall Officials: Daming Zhang, Study Director — Peking Union Medical College Hospital; Yikai Xu, Principal Investigator — Nanfang Hospital, Southern Medical University; Ting Liu, Study Director — First Affiliated Hospital Xi'an Jiaotong University
Locations (3):
- China (3):
  - Peking Union Medical College Hospital, Beijing
  - Nanfang Hospital, Guangzhou
  - The First Hospital of Xian Jiaotong University, Xi'an

IPD SHARING:
Plan to Share IPD: No